CLINICAL TRIAL: NCT06000085
Title: Clinical Performance of a Flowable Giomer Versus a Highly Viscous Glass-ionomer Cement in Restoring Class II Cavities of Primary Molars: A Randomized Clinical Trial
Brief Title: Clinical Performance of Two Different Restorative Materials in Restoring Class II Cavities of Primary Molars
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sarah Emad Ali El-Din, Assistant lecturer at the Pediatric Dentistry and Dental Public Health Department-Faculty of Dentistry, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PED 22-4D
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Dental Caries Class II
Keywords: proximal caries; primary molars; flowable giomer; equia forte

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flowable Giomer Beautifil flow plus x (Experimental): injectable flowable restorative material
  Interventions: Procedure: restoration of proximal cavities of primary molars with flowable giomer
- Glass-hybrid-added HVGIC Equia Forte (Active Comparator): Glass-hybrid-added Highly viscous glass ionomer cement
  Interventions: Procedure: restoration of proximal cavities of primary molars with highly viscous glass ionomer cement

INTERVENTIONS:
Procedure: restoration of proximal cavities of primary molars with flowable giomer — removal of proximal caries of primary molars and restoration of the cavities prepared by beautifil flow plus x
  Arms: Flowable Giomer Beautifil flow plus x
Procedure: restoration of proximal cavities of primary molars with highly viscous glass ionomer cement — removal of proximal caries of primary molars and restoration of the cavities prepared by equia forte
  Arms: Glass-hybrid-added HVGIC Equia Forte

SUMMARY:
The aim of the present study is to assess Flowable Giomer Beautifil Flow Plus X (Shofu Dental Corporation, Japan) and Glass-hybrid-added HVGIC, Equia Forte (GC Corporation, Tokyo,

Japan) in class II cavities of primary molars regarding the following objectives:

The primary objective To evaluate and compare the clinical performance of Flowable Giomer Beautifil Flow Plus X (Shofu Dental Corporation, Japan) and Glass-hybrid-added HVGIC, Equia Forte (GC Corporation, Tokyo, Japan) in restoring class II cavities of primary molars after 3,6, and 12 months. The secondary objective To assess the effect of different independent variables on the treatment outcome of the experimental restorative materials.

Research question:

Is there a difference in the clinical performance between flowable giomers and highly viscous glass ionomer in restoring class II cavities of primary molars?

Null Hypothesis There is no difference in the clinical performance between Flowable Giomer Beautifil Flow Plus X (Shofu Dental Corporation, Japan) and Glass-hybrid-added HVGIC, Equia Forte (GC Corporation, Tokyo, Japan) after one year of follow up.

DETAILED DESCRIPTION:
Study design:

The study will be two parallel-arm, double blinded randomized, controlled clinical trial with an equal allocation ratio.

Study Setting:

The study will be conducted at Pediatric dentistry and Dental Public Health Department, Faculty of Dentistry, Ain Shams University.

Ethical Considerations:

* The study methodology will be reviewed and approved by the faculty research ethical committee.
* Guardians of children will be asked to sign an informed consent in simple Arabic language before being enrolled in this study. The parents will be assured about confidentiality of all the collected data and were informed that their child has the right to withdraw at any given point during treatment without having to provide reasons for withdrawal.
* Children also will fill a simplified assent form.

Sample Size:

Sample size estimation was based on testing the null hypothesis that there is no difference between the clinical success rates of the two materials by setting α error of 5%, power of 80%, and allocation ratio 1:1. Results from previous studies suggested that the one-year clinical success rate of EQUIA Forte™ in class II restorations in primary molars was 74.4% (24) , while that for Beautifil flow plus x was estimated to be 94.1% based upon the findings of a previous study regarding Giomer in class II cavities. Based on this, the needed sample is 53 primary molars per group. Considering 15% drop-out rate, the needed sample size was increased to 62 molars per group. Sample size calculation was performed using G*Power software version 3.1.9.4 for MS Windows Study Population A total of 124 primary molars fulfilling the eligibility criteria will be restored in eligible participants, with one of the two tested restorative materials.

Study grouping:

The study will include two groups:

Group I (experimental): 62 primary molars will be restored with flowable Giomer beautifil flow plus x Group II (comparator): 62 primary molars will be restored with high-viscosity glass ionomer cement (EQUIA Forte)

Randomization and blinding:

Randomization will be performed using the Computer generated random number table to ensure that each primary molar had an equal chance of being assigned to either the glass ionomer group or the giomer group. Randomization will be done by tooth such that participants with multiple eligible carious primary molars were allowed to draw a corresponding number of cards. This trial will be double-blinded such that all participants, the clinical evaluator and the data analyst will be blinded to the type of the applied restorative materials in all periods of the study.

Allocation concealment:

The randomization groups will be written on a paper and each of the papers will be numbered and will be individually packed by another person than the investigator in an opaque envelope after folding each paper eight folds. All participants will be asked to select an opaque sealed envelope for each of their carious primary molars to avoid allocation bias. The numbers in the envelopes determined the group assigned for each molar. The investigator will open the sealed envelope after the cavity preparation and then assigns the treatment group accordingly.

Implementation:

A. Sequence generation will be done by a trial independent subject. B. Recruitment and screening of participants will be done by the main investigator, while enrolling of primary molars for the trial will be decided by two calibrated dentists.

Participants and assessors will be blinded at baseline and follow up. The primary investigator will not be blinded. C. Envelops will be kept with a trial independent subject and the allocated treatment will be revealed after cavity preparation

Study population:

Patients attending the Department of Pediatric Dentistry and dental public health, Faculty of Dentistry, at Ain Shams University for routine dental care will be examined clinically and radiographically with bite-wing radiography. Patients will be assessed for eligibility for participation.

Study Procedure

A detailed case history will be recorded, and an oral examination will be done. Oral prophylaxis will be performed to all the study children before the restorative treatment. A total of 124 primary molars (first/second, maxillary/mandibular) with carious lesions that indicated for restorative treatment will be selected by specified inclusion criteria. Based on the type of restorative material, the teeth will be randomly allocated to two groups (n = 62 in each group) Initial bite-wing radiographs of the teeth to be treated will be taken before the treatment.

Local anesthesia will be applied. Cavity preparations will be performed using diamond burs at high speed with water-cooling. Hand instruments and slow-speed tungsten carbide burs were used to remove the caries. Conservative cavity design will be used and beveling will not applied to the cavity walls to avoid unnecessary loss of hard dental tissue. The outline shape of the cavity will be limited to the removal of caries lesion. Any additional retention will not be prepared. The cavity will be rinsed and then dried with cotton pellets. A metal matrix band and wedges will be applied. Cotton rolls and a saliva ejector will be used for isolation.

Group 1 Giomer; Beautifil flow plus x After caries tissue removal, the cavity will be washed by rubbing wet cotton pellets against its walls to remove debris and remnants of decayed tissue removal. In the presence of the adjacent tooth, a matrix band and a wooden wedge were placed to adapt the restoration. A thin layer of the one-step self-etch adhesive BeautiBond (Shofu Inc) will be applied with a micro applicator and light cured for 10 s. The operator will place the Beautifil-flow plus x in increments creating the desired shape. Each increment will be light-cured for 20 s at each restoration surface. The composite will be used in increments up to 2 mm. An articulation paper will be used to check if there is any interference.

Group 2 Glass-hybrid-added HVGIC; Equia Forte:

The cavity will be conditioned with a poly- acrylic acid 'dentin conditioner' (EQUIA GC, JAPAN) which will be left for 15 seconds according to the manufacturer instructions. The conditioner will later be washed with a water spray, and then rinsing water will be blotted with a dry cotton pellet, leaving a moist surface. Each capsule of high viscous glass ionomer cement will be mixed for 10 seconds using amalgamator according to the manufacturer's instructions then packed into the prepared cavity with a carver and ball burnisher. Any excess material will be removed using a carver. Finally, a thin layer of the Equia Forte Coat ® (GC Corp) will be applied with a micro applicator and then light-cured for 20 s. An articulation paper will be used to check if the restoration caused any occlusal interference.

ELIGIBILITY:
Inclusion Criteria:

inclusion criteria of study participants:

1. 4 to 8 years old medically free children.
2. Cooperative children classified as class 3 or 4 based on Frankel et al. classification
3. Children who had at least one active dentinal carious lesion on proximal surface of primary molars

inclusion criteria of teeth:

1. Primary molars with active dentinal carious lesion on their proximal surface score 4, 5 using ICDAS.
2. Primary molars with proximal carious lesion extended to outer and middle third of dentin scored D1and D2 that will be detected by bitewing radiograph.
3. Simple or compound class II cavities be present
4. The antagonist and the adjacent tooth should be present
5. Primary molar should have at least 2/3 of the root present

Exclusion Criteria:

exclusion criteria of study participants

1. Refusal of the parents to sign the informed consent
2. Presence of deep bite or any pictures of malocclusion and any parafunctional habits.

exclusion criteria of teeth

1. Presence of any unprovoked pain, pulp exposure,clinical swelling, abscess or fistula.
2. Presence of any physiological or pathological mobility.
3. Very deep subgingival cavities
4. Teeth with congenitally missing successor

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 124 (Estimated)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
The clinical performance of Flowable Giomer Beautifil Flow Plus X (Shofu Dental Corporation, Japan) and Glass-hybrid-added HVGIC, Equia Forte (GC Corporation, Tokyo, Japan) in restoring class II cavities of primary molars | 12 months
  The restorations will be evaluated using the FDI criteria having esthetic, functional, and biological properties

SECONDARY OUTCOMES:
The effect of different independent variables on the treatment outcome of the experimental restorative materials. | 12 months
  assessment of the effect of different variables such as the age of the patient and the properties of the tooth on the restoration survival

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Emad, Principal Investigator — faculty of dentistry ain shams university
Locations (1):
- Faculty of dentistry ain shams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No